CLINICAL TRIAL: NCT06386250
Title: Comparison of Regional Block, Caudal Block and Wound Infiltration for Post-operative Pain Management in Children Undergoing Inguinal Herniotomy
Brief Title: Comparison of Regional Block, Caudal Block and Wound Infiltration in Inguinal Hernitomy
Acronym: Painseverity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Edward Medical University (Other)
Responsible Party: Principal Investigator, Muhammad Sharif, PROFESSOR, King Edward Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0005
Record Dates: First submitted 2024-04-13; First posted 2024-04-26 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Postoperative Pain
Keywords: Postoperative pain; inguinal herniotomy; children; regional block; caudal block; wound infilteration
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine; Injections, Epidural

STUDY DESIGN:
Intervention Model Description: Regional block group (Group A), wound infiltration group (Group B), caudal block group (Group C)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Active Comparator): In group A, iliohypogastric and ilioinguinal nerves were blocked by using 0.25% bupivacaine 2ml/kg of combined with skin infiltration of adrenaline 1:200 000.
  Interventions: Procedure: regional block; Procedure: Caudal block; Procedure: Epidural
- Group B (Active Comparator): In group B 0.25% bupivacaine 0.5ml/Kg was infiltrated at the surgical site.
  Interventions: Procedure: regional block; Procedure: Caudal block; Procedure: Epidural
- Group C (Experimental): In group C 0.25% Bupivacaine 1ml /kg was given into epidural space at L4-L5 or L5-S1.
  Interventions: Procedure: regional block; Procedure: Caudal block; Procedure: Epidural

INTERVENTIONS:
Procedure: regional block — In group A, iliohypogastric and ilioinguinal nerves were blocked by using 0.25% bupivacaine 2ml/kg of combined with skin infiltration of adrenaline 1:200 000.
  Other Names: wound infilteration
Procedure: Caudal block — In group B 0.25% bupivacaine 0.5ml/Kg was infiltrated at the surgical site.
  Other Names: infilteration with 0.25% bupivacaine
Procedure: Epidural — In group C 0.25% Bupivacaine 1ml /kg was given into epidural space at L4-L5 or L5-S1.
  Other Names: injection Bupivacaine into epidural space

SUMMARY:
Background: Although Inguinal herniotomy in children is taken as a day care procedure, post-operative pain management still remain controversial in these cases and superiority of wound infiltration, caudal block or regional block over each isn't known.

Objective: The objective of the study was compare regional block, caudal block and wound infiltration for post-operative pain management in children undergoing inguinal herniotomy

DETAILED DESCRIPTION:
Three hundred patients rom the department of pediatric surgery, KEMU/Mayo Hospital, were randomized in three study groups by a computer generated table. Regional block group (Group A), wound infiltration group (Group B), caudal block group (Group C). . Patients were assessed for postoperative pain intensity using FLACC pain scale at 0, 1, 2, 4, 8, 24 hours after surgery in children less than 8 years of age. Wong-Baker Faces pain Scale at 0, 1, 2, 4, 8, 24 hours after surgery in children more than 8 years of age. Patients were discharged after 24 hours. If pain score ≥ 4 was given intravenously, Ketoralac. Urinary retention was observed after 24 hours, wound infection was observed after 7 days.

ELIGIBILITY:
Inclusion Criteria:

* Both Male and female inguinal hernia patients
* Patients from 3-12 years age Exclusion Criteria
* History of allergy to any drugs used in study documented on history .Infection at the site of regional, caudal or local infiltration, documented on clinical examination.

.Irreducible, obstructed or strangulated hernia, documented on clinical examination.

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 300 (Actual)
Dates: Start 2019-01-05 (Actual); Primary Completion 2020-01-06 (Actual); Study Completion 2020-01-06 (Actual)

PRIMARY OUTCOMES:
Postoperative pain intensity | 24 hours
  Patients were assessed for postoperative pain intensity using FLACC pain scale at 0, 1, 2, 4, 8, 24 hours after surgery in children less than 8 years of age. Wong-Baker Faces pain Scale at 0, 1, 2, 4, 8, 24 hours after surgery in children more than 8 years of age.

OTHER OUTCOMES:
postoperative pain intesity | 24 hours
  Wong-Baker Faces pain Scale at 0, 1, 2, 4, 8, 24 hours after surgery in children more than 8 years of age.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Sharif, FCPS, Study Chair — King edward Medical University/Mayo Hospital Lahore
Locations (1):
- Muhammad Sharif, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
will be shared on request